CLINICAL TRIAL: NCT01802879
Title: An Open-label Multi-center Single Agent Panobinostat Roll-over Protocol for Patients Who Have Completed a Previous Novartis-sponsored Panobinostat Study and Are Judged by the Investigator to Benefit From Continued Single Agent Panobinostat Treatment
Brief Title: Study to Allow Access to Single Agent Panobinostat for Patients Who Are on s.a. Panobinostat Treatment in a Novartis-sponsored Study and Continue to Benefit From the Treatment as Judged by the Investigator
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLBH589B2402B; 2012-005252-41 (EudraCT Number)
Record Dates: First submitted 2013-02-26; First posted 2013-03-04 (Estimated); Results first posted 2019-12-06 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-11

CONDITIONS: Hematologic Neoplasms
Keywords: Hematologic Neoplasms, LBH589,; Panobinostat,
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Panobinostat - 10 to 40 mg/day TIW QoW (Experimental): 10 to 40mg/day TIW QoW (3 times/week every other week) as per parent protocol design
  Interventions: Drug: Panobinostat

INTERVENTIONS:
Drug: Panobinostat — Panobinostat was provided as 5, 10 and 20 mg hard gelatin capsules to be taken orally. Patients started on dose from parent protocol and dose modifications were at the discretion of the investigator based on guidance provided in the protocol and IB.

SUMMARY:
The study allowed continued use of single agent panobinostat in patients who were on single agent panobinostat treatment in a Novartis-sponsored study which had met its endpoint and were benefiting from the treatment as judged by the investigator.

DETAILED DESCRIPTION:
This was a multi-center open label study to provide continued use of single agent oral panobinostat to patients treated in a Novartis-sponsored study (parent study) which had met its endpoint and were benefiting from continuation of the treatment with single-agent panobinostat as judged by the investigator. Patients from multiple parent studies were transferred over to this protocol and continued to receive single agent panobinostat at the last assigned dose and regimen of the parent protocol. There was no screening period, and patients had to visit the study center at least on a quarterly basis. During these visits limited information on study treatment and occurrence of SAEs was collected for the clinical database. SAEs were only reported to the Novartis safety database. Other assessments and possibly more frequent visits occurred as per standard of care at the site. Patients continued treatment until they were no longer benefiting from panobinostat treatment, developed unacceptable toxicities, withdrew consent, were non-compliant with the protocol, the investigator believed it was no longer in the best interest to continue, the patient died, or for other administrative reasons. An end of treatment visit and a safety follow-up for 30 days after the last dose was performed. The study was expected to remain open for 5 years or until such time that enrolled patients no longer needed treatment with panobinostat, whichever came earlier.

ELIGIBILITY:
Inclusion Criteria:

* patient had been enrolled in a Novartis-sponsored, Oncology OGD&GMA study receiving s.a. oral panobinostat and had fulfilled all their requirements in the parent study
* patient had been benefiting from the treatment with s.a. oral panobinostat as determined by the guidelines of the parent protocol and according to the Investigator's clinical judgment
* patient had demonstated compliance
* patient had given written informed consent.

Exclusion Criteria:

* patient had been permanently discontinued from s.a. oral panobinostat study treatment in the parent study due to unacceptable toxicity, withdrawal of consent, non-compliance to study procedures or any other reason (including progression of disease).
* patient had participated in a Novartis sponsored combincation trial where panobinostat was dispensed in combination with another study medication and was still receiving combination therapy
* patient was pregnant or nursing at the time of entry
* women of child-bearing potential and male patients with sexual partners of child-bearing potential who were unwilling to use highly effective methods of contraception during dosing and for a specified duration after stopping study treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-06-24 (Actual); Primary Completion 2018-11-19 (Actual); Study Completion 2018-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- United States (4):
  - City of Hope National Medical Center Dept.ofCityofHopeMedicalCtr(1), Duarte, California
  - Georgia Regents University SC-2, Augusta, Georgia
  - Dana Farber Cancer Institute Reg. Ped, Boston, Massachusetts
  - University of Utah / Huntsman Cancer Institute SC-2, Salt Lake City, Utah
- Novartis Investigative Site, Jerusalem, Israel
- Novartis Investigative Site, Leiden, Netherlands
- Novartis Investigative Site, Salamanca, Castille and León, Spain

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There was no screening period. Patients enrolled into trial directly from the parent protocol.
Period: Overall Study
Arm/Group | Panobinostat - 10 to 40 mg/Day TIW QoW
Started | 8
Completed | 0
Not Completed | 8
Not completed — Administrative problems | 2
Not completed — Disease progression | 6

BASELINE CHARACTERISTICS:
Arm/Group | Panobinostat - 10 to 40 mg/Day TIW QoW
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Parent protocol participants [Number; unit: participants]
  CLBH589B2201 | 2
  CLBH589B2207 | 3
  CLBH589E2214 | 1
  CLBH589X2105 | 2

OUTCOME MEASURES:

1. Secondary Outcome: Percentage of Patients With Clinical Benefit as Assessed by the Investigator.
Description: Patients were assessed by investigators at scheduled visits to determine if patient continued to benefit from panobinostat therapy.
Time Frame: baseline up to approximate 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Panobinostat - 10 to 40 mg/Day TIW QoW
Number analyzed (Participants) | 8
Participants
  Participants with clinical benefit | 7

2. Primary Outcome: Overview of Adverse Events (Safety Set)
Description: Adverse events were collected from baseline up to 30 days post treatment at scheduled visits. Severity of adverse events was assessed according to the current version of Common Terminology Criteria for Adverse Events (CTCAE). If CTCAE grading did not exist for an adverse event, the severity of mild, moderate, severe, and life-threatening, corresponding to Grades 1 - 4, was used
Time Frame: Baseline up to approximately 60 months
Measure: Number; unit: participants
Arm/Group | Panobinostat - 10 to 40 mg/Day TIW QoW
Number analyzed (Participants) | 8
participants
  Any adverse event (AE) | 6
  Any treatment related AE | 2
  Any serious adverse event (SAE) | 2
  Grade 3 or 4 AE | 3
  Grade 3 or 4 AE - suspected to be related | 1
  AEs leading discontinuation | 0
  AEs leading to dose adjust/ temp dose interruption | 2
  On-treatment death | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment plus 30 days post treatment, up to maximum duration of 84 weeks
Description: AE additional description
Arm/Group | Panobinostat - 10 to 40 mg/Day TIW QoW
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 2/8
Other Adverse Events (participants affected / at risk) | 4/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Panobinostat - 10 to 40 mg/Day TIW QoW (N=8)
Non-cardiac chest pain (General disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Panobinostat - 10 to 40 mg/Day TIW QoW (N=8)
Neutropenia (Blood and lymphatic system disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Gastric disorder (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Nasopharyngitis (Infections and infestations) | 1
Blood creatinine increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Benign muscle neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neuropathy peripheral (Nervous system disorders) | 2
Insomnia (Psychiatric disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-03-11): https://cdn.clinicaltrials.gov/large-docs/79/NCT01802879/Prot_000.pdf
  • Statistical Analysis Plan (2016-06-14): https://cdn.clinicaltrials.gov/large-docs/79/NCT01802879/SAP_001.pdf